CLINICAL TRIAL: NCT06306690
Title: Biomarkers for Prognosis in Different Forms of Retinitis Pigmentosa
Brief Title: Biomarkers in Retinitis Pigmentosa
Acronym: RPMARKER
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RIZZO STANISLAO, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6401
Record Dates: First submitted 2024-02-10; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; Retinal degeneration; Multimodal imaging; electroretinography; retinal pigment epithelium and outer retinal atrophy (RORA)
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Degeneration | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 1. Patients with rhodopsin mutation (RHO): Following a clinical diagnosis, patients undergo genetic testing. Patients with rhodopsin mutation (RHO) a mutation are categorised into subgroup 1.
  Interventions: Diagnostic Test: OCT, OCT angiography, flicker ERG and Ultra Wide Field retinography and autofluorescence.
- 2. Patients with pre-mRNA factor 8 (PRPF8) mutation: Following a clinical diagnosis, patients undergo genetic testing. Patients with pre-mRNA factor 8 (PRPF8) mutation are categorised into subgroup 2.
  Interventions: Diagnostic Test: OCT, OCT angiography, flicker ERG and Ultra Wide Field retinography and autofluorescence.
- 3.Patients a cone-specific phosphodiesterase, i.e. PDE6B, mutation: Following a clinical diagnosis, patients undergo genetic testing. Patients with a cone-specific phosphodiesterase, i.e. PDE6B, mutation are categorised into subgroup 3.
  Interventions: Diagnostic Test: OCT, OCT angiography, flicker ERG and Ultra Wide Field retinography and autofluorescence.
- 4. Patients with Chromosome 2-Open (C2orf71) mutation: Following a clinical diagnosis, patients undergo genetic testing. Patients with Chromosome 2-Open (C2orf71) mutation are categorised into subgroup 4.
  Interventions: Diagnostic Test: OCT, OCT angiography, flicker ERG and Ultra Wide Field retinography and autofluorescence.
- 5. Patients with Guanylate Cyclase (GUCY2D) mutation: Following a clinical diagnosis, patients undergo genetic testing. Patients with Guanylate Cyclase (GUCY2D) mutation are categorised into subgroup 5.
  Interventions: Diagnostic Test: OCT, OCT angiography, flicker ERG and Ultra Wide Field retinography and autofluorescence.
- 6. Patients with RP- specific nuclear receptor (Nr2E3) mutation: Following a clinical diagnosis, patients undergo genetic testing. Patients with RP- specific nuclear receptor (Nr2E3) mutation are categorised into subgroup 6.
  Interventions: Diagnostic Test: OCT, OCT angiography, flicker ERG and Ultra Wide Field retinography and autofluorescence.

INTERVENTIONS:
Diagnostic Test: OCT, OCT angiography, flicker ERG and Ultra Wide Field retinography and autofluorescence. — the best visual acuity will be evaluated using decimal tables and then converted to logMar.
  Ocular fundus examination will be evaluated following pharmacological mydriasis with Tropicamide 1%.
  OCT will be essential to quantify the central macular thickness and the thickness of the RPE.
  OCT angiography is a non-invasive method to assess the presence or absence of neovascular membrane and macular flow density.
  Color and ultra wide field autofluorescence images of the retina will be performed with Zeiss Clarus retinography to search for signs that identify different types of RP and predict their activity and evolution.
  Electroretinogram flicker (ERG) is a common measure of cone pathway function that is used to study the normal visual system and that of patients with inherited and acquired retinal dysfunction Measurements will be performed using an electrophysiological recording system (CSO). Intermittent stimuli are presented using a Ganzfeld dome (CSO).

SUMMARY:
The objective of this study is to discover biomarkers that demonstrate a correlation between the severity of retinitis pigmentosa (RP) and the thickness of the retinal pigment epithelium (RPE). These biomarkers will serve as prognostic indicators for various kinds of retinitis pigmentosa. The objective of this study is to find biomarkers that establish a correlation between the severity of retinitis pigmentosa and the thickness of the retinal pigment epithelium (RPE), which can serve as a prognostic indicator for Retinitis Pigmentosa.

DETAILED DESCRIPTION:
After a genetic confirmation of RP and classification, the patients will undergo a comprehensive ophthalmological examination that includes the following tests: slit-lamp anterior segment, visual acuity direct and indirect ophthalmoscopy, intraocular pressure, and family history.In order to evaluate the potential role of RPE in the advancement of RP, HD-OCT and OCT angiography images of the outer retina using OCT devices will be performed.

Analysis of high-resolution images captured with an ultrawidefield system using a Zeiss Clarus device in order to determine the condition of the peripheral retina.Finally, Flicker Electroretinogram (fERG) performed on the central retina (macula), to assess the central macular function within an 18° field of view. This assessment involved measuring the response of the macula to a flickering stimulus with a frequency of 41 Hz, which is commonly done in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to read and sign informed consent
* Patients with Retinitis pigmentosa confirmed by genetic test.
* Patients older than or equal to 18 years of age

Exclusion Criteria:

* Other retinal diseases such as macular hole, retinal detachment, macular neovascularization.
* Corneal surgery in the last 12 months
* Glaucoma with pressure above 25 mmHg in the last three months.
* Best Correct Visual Acuity below 1/10 in at least one eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be enrolled at the Ophthalmology department of Fondazione Policlinico Universitario A. Gemelli IRCCS.
  Patients with diverse kinds of RP with genetic confirmation, no other retinal disorders, pressure under 25 mmHg for three months, and no corneal surgery in the past year are included.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Retinal pigment epithelium changes in Retinitis Pigmentosa. | 14 months
  Retinal pigment epithelium extent measured with OCT calliper (micrometers).

SECONDARY OUTCOMES:
Retinitis Pigmentosa biomarkers | 14 months
  Measurement of retinal pigment epithelium extension by oct calliper (micrometers) in different forms of retinitis pigmentosa.
  Measurement of superficial and deep retinal vascularisation in the different forms of retinitis pigmentosa.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Cristina Savastano, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Campochiaro PA, Mir TA. The mechanism of cone cell death in Retinitis Pigmentosa. Prog Retin Eye Res. 2018 Jan;62:24-37. doi: 10.1016/j.preteyeres.2017.08.004. Epub 2017 Sep 27. PMID 28962928
- [Background] Dias MF, Joo K, Kemp JA, Fialho SL, da Silva Cunha A Jr, Woo SJ, Kwon YJ. Molecular genetics and emerging therapies for retinitis pigmentosa: Basic research and clinical perspectives. Prog Retin Eye Res. 2018 Mar;63:107-131. doi: 10.1016/j.preteyeres.2017.10.004. Epub 2017 Oct 31. PMID 29097191
- [Background] Cross N, van Steen C, Zegaoui Y, Satherley A, Angelillo L. Retinitis Pigmentosa: Burden of Disease and Current Unmet Needs. Clin Ophthalmol. 2022 Jun 20;16:1993-2010. doi: 10.2147/OPTH.S365486. eCollection 2022. PMID 35757022
- [Background] Chaumet-Riffaud AE, Chaumet-Riffaud P, Cariou A, Devisme C, Audo I, Sahel JA, Mohand-Said S. Impact of Retinitis Pigmentosa on Quality of Life, Mental Health, and Employment Among Young Adults. Am J Ophthalmol. 2017 May;177:169-174. doi: 10.1016/j.ajo.2017.02.016. Epub 2017 Feb 22. PMID 28237413
- [Background] Hartong DT, Berson EL, Dryja TP. Retinitis pigmentosa. Lancet. 2006 Nov 18;368(9549):1795-809. doi: 10.1016/S0140-6736(06)69740-7. PMID 17113430
- [Background] Wu KY, Kulbay M, Toameh D, Xu AQ, Kalevar A, Tran SD. Retinitis Pigmentosa: Novel Therapeutic Targets and Drug Development. Pharmaceutics. 2023 Feb 17;15(2):685. doi: 10.3390/pharmaceutics15020685. PMID 36840007
- [Background] Russell S, Bennett J, Wellman JA, Chung DC, Yu ZF, Tillman A, Wittes J, Pappas J, Elci O, McCague S, Cross D, Marshall KA, Walshire J, Kehoe TL, Reichert H, Davis M, Raffini L, George LA, Hudson FP, Dingfield L, Zhu X, Haller JA, Sohn EH, Mahajan VB, Pfeifer W, Weckmann M, Johnson C, Gewaily D, Drack A, Stone E, Wachtel K, Simonelli F, Leroy BP, Wright JF, High KA, Maguire AM. Efficacy and safety of voretigene neparvovec (AAV2-hRPE65v2) in patients with RPE65-mediated inherited retinal dystrophy: a randomised, controlled, open-label, phase 3 trial. Lancet. 2017 Aug 26;390(10097):849-860. doi: 10.1016/S0140-6736(17)31868-8. Epub 2017 Jul 14. PMID 28712537
- [Background] Iftikhar M, Lemus M, Usmani B, Campochiaro PA, Sahel JA, Scholl HPN, Shah SMA. Classification of disease severity in retinitis pigmentosa. Br J Ophthalmol. 2019 Nov;103(11):1595-1599. doi: 10.1136/bjophthalmol-2018-313669. Epub 2019 Jan 31. PMID 30705041
- [Background] Savastano MC, Falsini B, Ferrara S, Scampoli A, Piccardi M, Savastano A, Rizzo S. Subretinal Pigment Epithelium Illumination Combined With Focal Electroretinogram and Visual Acuity for Early Diagnosis and Prognosis of Non-Exudative Age-Related Macular Degeneration: New Insights for Personalized Medicine. Transl Vis Sci Technol. 2022 Jan 3;11(1):35. doi: 10.1167/tvst.11.1.35. PMID 35077530
- [Background] Guymer RH, Rosenfeld PJ, Curcio CA, Holz FG, Staurenghi G, Freund KB, Schmitz-Valckenberg S, Sparrow J, Spaide RF, Tufail A, Chakravarthy U, Jaffe GJ, Csaky K, Sarraf D, Mones JM, Tadayoni R, Grunwald J, Bottoni F, Liakopoulos S, Pauleikhoff D, Pagliarini S, Chew EY, Viola F, Fleckenstein M, Blodi BA, Lim TH, Chong V, Lutty J, Bird AC, Sadda SR. Incomplete Retinal Pigment Epithelial and Outer Retinal Atrophy in Age-Related Macular Degeneration: Classification of Atrophy Meeting Report 4. Ophthalmology. 2020 Mar;127(3):394-409. doi: 10.1016/j.ophtha.2019.09.035. Epub 2019 Sep 30. PMID 31708275
- [Background] Placidi G, Maltese PE, Savastano MC, D'Agostino E, Cestrone V, Bertelli M, Chiurazzi P, Maceroni M, Minnella AM, Ziccardi L, Parisi V, Rizzo S, Falsini B. Retinitis Pigmentosa Associated with EYS Gene Mutations: Disease Severity Staging and Central Retina Atrophy. Diagnostics (Basel). 2023 Feb 23;13(5):850. doi: 10.3390/diagnostics13050850. PMID 36899994